CLINICAL TRIAL: NCT06260215
Title: Recovery Kinetics Following a Soccer Training in Middle-aged Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FFH
Record Dates: First submitted 2024-01-29; First posted 2024-02-15 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2024-02

CONDITIONS: Skeletal Muscle Damage
Keywords: Recovery; Soccer; Soccer training; performance; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in this arm will receive no intervention
- SoccerTraining (Experimental): Participants in this arm will participate in a soccer training (ST) session for 60 minutes. During the training the participans will execute the warm-up process, the part of soccer technical exercises and they will play a small-side-game.
  Interventions: Other: ST

INTERVENTIONS:
Other: ST — Participants will perform a soccer training (ST) session for 60 minutes. The training will include the warm-up, soccer technical exercises and a small-side game
  Arms: SoccerTraining

SUMMARY:
This study aims at investigating the recovery kinetics of skeletal muscle damage, neuromuscular fatigue and performance following a single soccer trainning session in middle aged males. The participants will perform a soccer training session [A single training session including 60 minutes of warm up, soccer technical exercises and small-sided game] and a cotrol trial (No intervention included, only daily measurements) in randomized, repeated measures, crossover design. Assesesments related to skeletal muscle damage, performance and neuromuscular fatigue will be executed before the training session and daily for four consecutive days after training.

DETAILED DESCRIPTION:
Eleven male middle-aged participants will be included in this study. Participants will be initially informed about the main goals of study as well as the associated risks and benefits and then will provide their signed consent form. At baseline, they will undergo assessment of their anthropometrics (body mass, height, BMI, WHR), body compotition (using DXA), physical contition level (peak oxygen consumption, VO2peak), haemodynamic profile (diastolic and diastolic blood pressure) and daily dietary intake.Thereafter, they will participate in two experimental trials (Control trial and Soccer trial) in a randomized, crossover, repeated measure design: 1) ST (Soccer Trial): Participants in this trial will perform a soccer training session (60 min) consisted of warm-up, technical exercises and small-sided game, CT (Control Trial): Participants in this trial will only execute the evaluations daily in the dependent variables (they will not receive any intervention). Before each trial, the participants will provide a resting blood sample (for the determination of white blood cells, granulocyte cells, monocyte cells, lymphocyte cells, Hemeatocrit, Hemoglobin, red blood cells and platelets, total antioxidant capacity, glutathione and creatine kinase activity) and undergo assessments of their delay onset muscle soreness (DOMS), maximal voluntary isometric contraction (MVIC) of knee extensors and flexors (by isokinetic dynamometer), height and power of countermovement jump (CMJ-using force platform), 10m and 30m sprint time (will be evaluated using light cells). A 7-day wash-out period will apllied between ST and CT. The blood sample will be collected before and 24, 48 and 72 hours post-taining. Also, the evaluation of DOMS, MVIC, sprinting performance, power and jump height (by CMJ) will be evaluated before and 24, 48, 72 and 96 hours post training.

ELIGIBILITY:
Inclusion Criteria:

* Free of musculoskeletal injuries
* No use of ergogenic supplements or medication
* Free of chronic diseases
* age of 40-60 years

Exclusion Criteria:

* Musculoskeletal injury
* Use of alcohol, caffeine and any type of ergogenic supplements or medication during the course of the study

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-03-09 (Actual)

PRIMARY OUTCOMES:
Change in White blood cell count | At baseline, at 24, 48 and 72 hours after soccer training
  White blood cell count will be measured using an automatic blood analyzer
Change in Granulocyte cell count | At baseline, at 24, 48 and 72 hours after soccer training
  Change in White blood cell count will be measured using an automatic blood analyzer
Change in Platelets cell count | At baseline, at 24, 48 and 72 hours after soccer training
  Platelets cell count will be measured using an automatic blood analyzer
Change in Monocyte cell count | At baseline, at 24, 48 and 72 hours after soccer training
  Monocytes cell count will be measured using an automatic blood analyzer
Change in Lymphocyte cell count | At baseline, at 24, 48 and 72 hours after soccer training
  Lymphocyte cell count will be measured using an automatic blood analyzer
Change in percentage of Hematocrit level | At baseline, at 24, 48 and 72 hours after soccer training
  The percentage of Hematocrit level will be measured using an automatic blood analyzer
Change Red blood cells count | At baseline, at 24, 48 and 72 hours after soccer training
  Red blood cells count will be measured using an automatic blood analyzer
Change in Hemoglobin level | At baseline, at 24, 48 and 72 hours after soccer training
  Hemoglobin level will be measured using an automatic blood analyzer
Change in Creatine kinase activity | At baseline, at 24, 48 and 72 hours after soccer training
  Creatine kinase activity will be measured in plasma
Change in Total antioxidant capacity | At baseline, at 24, 48 and 72 hours after soccer training
  Total antioxidant capacity will be measured in plasma
Change in Glutathione concentration in blood | At baseline, at 24, 48 and 72 hours after soccer training
  Glutathione concentration will be measured in red blood cells
Change in countermovement jump height | At baseline, at 24, 48, 72 and 96 hours after soccer training
  countermovement jump height will be measured using a force platform
Change in Peak power during coutermovement jump test | At baseline, at 24, 48, 72 and 96 hours after soccer training
  The peak power will be measured using a force platform
Change in isometric peak torque of knee extensors and flexors | At baseline, at 24, 48, 72 and 96 hours after soccer training
  Isometric peak torque will be assessed on an isokinetic dynamometer
Change in sprint time of 10 m | At baseline, at 24, 48, 72 and 96 hours after soccer training
  10m sprint time will be assessed using light cells
Change in sprint time of 30 m | At baseline, at 24, 48, 72 and 96 hours after soccer training
  30m sprint time will be assessed using light cells
Change in delayed onset of muscle soreness | At baseline, at 24, 48, 72 and 96 hours after soccer training
  Muscle soreness will be assessed by palpation of muscle belly and the distal region

SECONDARY OUTCOMES:
Dietary intake | At baseline
  Dietary intake will be assesed over a 7-day period using diet recalls
Peak Maximal oxygen consumption (Peak VO2) | At baseline
  Peak VO2 will be estimated by open circuit spirometry via breath by breath method
Body Mass | At baseline
  Body Mass will be measured on a beam balance with stadiometer
Body Height | At baseline
  Body Height will be measured on a beam balance with stadiometer
Body Fat | At baseline
  Body Fat will be measured by using Dual-emission X-ray absorptiometry
Lean body mass | At baseline
  Lean body mass will be measured by using Dual-emission X-ray absorptiometry
Bone mass density | At baseline
  Bone mass density will be measured by using Dual-emission X-ray absorptiometry
Bone mass content | At baseline
  Bone mass content will be measured by using Dual-emission X-ray absorptiometry
Field activity during the soccer training | During the 60 minutes soccer training (ST) session (72 hours after baseline measurements)
  The field activity will be continuously monitored during the soccer training using global positioning system (GPS)
Heart rate during the soccer training | During the 60 minutes soccer training (ST) session (72 hours after baseline measurements)
  Heart rate will be continuously monitored during the soccer training using heart rate monitors
Systolic Blood Pressure | At baseline
  Systolic Blood Pressure will be examined using sphygmomanometer
Dystolic Blood Pressure | At baseline
  Dystolic Blood Pressure will be examined using sphygmomanometer
Rest Heart Rate | At baseline
  The rest heart rate will be estimated using a heart rate monitor

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis G Fatouros, Prof, Study Director — University of Thessaly
Locations (1):
- University o Thessaly, School of Physical Education and Sports Science, Trikala, Greece